CLINICAL TRIAL: NCT04466774
Title: A Comparative, Controlled Study to Evaluate the Lay User Accuracy and Performance of the Dip Home-Based Dipstick Analyzer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Healthy.io Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTP-Healthy.io-01
Record Dates: First submitted 2020-07-01; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Urine Detectable Acute and Chronic Diseases
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Dip Home-Based Dipstick Analyzer (Experimental): Each participant will test their urine sample using the HBDA. device
  Interventions: Diagnostic Test: Dip Home-Based Dipstick Analyzer; Device: Urine analysis predicate device for professional user

INTERVENTIONS:
Diagnostic Test: Dip Home-Based Dipstick Analyzer — The Dip Home-Based Dipstick Analyzer is a prescription, in-vitro diagnostic, home use device, which qualitatively and semi-quantitatively measures six urine analytes. The device combines a urine stick kit with an easy to use smartphone application using an image recognition algorithm.
Device: Urine analysis predicate device for professional user — Results of the experimental HBDA device will be compared to the results of the predicate device tested by a professional user.

SUMMARY:
The Dip Home-Based Dipstick Analyzer (henceforth HBDA) is composed of a kit and a smartphone application. The device will be provided to the subject in a simulated home-use environment. All subjects will be asked to complete the urine test by following the application guidance, including providing a urine sample and scanning the urine strip after placing it on the Color-Board.

The user will also complete a questionnaire to collect information regarding the use of the HBDA device. Following the usability test performed by the lay user, the subject's urine sample will be tested by the professional user using the comparator device. The use of the HBDA device will be evaluated for accuracy and identified risks. Additionally, measurable usability criteria for specific, critical steps will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-80 years of age
* Subjects who are healthy or pregnant; or
* Subjects diagnosed with a disease that normally represents itself with an abnormal concentration of one of the following urine analytes; Glucose, Bilirubin, Ketone (Acetoacetic acid), Specific Gravity, Blood, pH, Protein, Urobilinogen, Leukocytes, and Nitrite
* Subject is capable and willing to provide informed consent.
* Subject has facility with both hands.
* Subject is capable and willing to adhere to the study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 429 (Actual)
Dates: Start 2017-03-05 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of the % agreement of the Dip HBDA, tested by the lay user, as compared to a comparator device, tested by a professional user. | 11 months

SECONDARY OUTCOMES:
Evaluation of the Dip HBDA usability success rate, by potential lay users under actual use conditions. | 11 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Activmed Practices & Research, Inc., Methuen, Massachusetts
  - AccuMed research associates, Garden City, New York